CLINICAL TRIAL: NCT01784289
Title: Adipocyte, Insulin-resistance and Immunity : Evaluation of Interleukin-7 in Lipodystrophies According to Fat Mass and Glucose Metabolism
Brief Title: Adipocyte, Insulin-resistance and Immunity : Evaluation of Interleukin-7 in Lipodystrophy, Diabetes and Obesity
Acronym: IL-7norm
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_09/0941; 2009-A01169-48 (Other: ID-RCB number, ANSM); B91413-80 (Other: AFSSAPS); PHRC 2009/API (Other: DHOS)
Record Dates: First submitted 2011-08-09; First posted 2013-02-05 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Lipodystrophy; Obesity; Type 2 Diabetes
Keywords: Interleukin 7; adipose tissue
MeSH Terms: conditions — Lipodystrophy; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Wholeblood and tissue bank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- normal: Patients with no overweight and no type 2 diabetes
- lipodystrophy: patients with a lipodystrophy, most are diabetics
- obese non diabetics: Patients with obesity (BMI <30kg/m2), without diabetes
- obese diabetics: Patients with obesity (BMI <30 kg/m2), with diabetes

SUMMARY:
White adipose tissue-related diseases spread from excess (obesity) to lack (lipoatrophies) through aberrant distribution (lipodystrophies), these 3 different disorders being paradoxically able to induce a metabolic insulin resistance syndrome. The respective part of quantitative and qualitative anomalies of adipose tissue, gluco- and lipo-toxicity, liver and muscle insulin resistance, low-grade fat inflammation and immune alterations are not perfectly understood in the metabolic syndrome yet. Therefore, the aim of this study is to assess different cytokines, especially interleukin 7, and metabolic parameters as well as fat mass distribution with DEXA and RMN, in different models of fat distribution, including normal-weight, obese and lipodystrophic patients. A plasma serum, gene and adipose tissue bank will be constituted at the same time to improve our knowledge in disorders linking fat mass, insulin resistance and immunity, especially in lipodystrophies, a rare monogenic model of insulin resistance.

DETAILED DESCRIPTION:
Rational: In reason of its ability to store fatty acids and to secrete numerous pro-inflammatory cytokines, the adipocyte appears as a key cell in the regulation of energy metabolism and immune response. Moreover, it has been recently shown that adipocytes play a role in the recruitment of cells involved in innate and adaptive immunity in adipose tissue.

White adipose tissue-related diseases are numerous, spreading from excess (obesity) to a complete (lipoatrophies) or partial lack (lipodystrophies), these 3 different disorders being paradoxically able to induce a metabolic insulin resistance syndrome.

Among the involved cytokines, interleukin-7 (IL-7), mostly known for its immune functions, also participates to the quantitative and qualitative balance of fat mass. Thus, IL-7 over-expression in an animal model induces a lipodystrophic syndrome with insulin resistance whereas in humans, a preliminary study shows that LMNA-linked lipodystrophies are associated with an increase of blood IL-7 levels. IL-7 also participates to reactivation of autoimmunity in patients suffering from auto-immune type 1 after islet transplantation.

Therefore, the aim of this study is to assess different cytokines, especially interleukin 7, and metabolic parameters levels as well as fat mass distribution, in different models of fat distribution, including normal-weighed, obese and lipodystrophic patients. A plasma serum, gene and tissue bank will be constituted in order to improve our knowledge in disorders linking fat mass, insulin resistance and immunity, especially in lipodystrophies, a rare monogenic model of insulin resistance.

Patients: The included patients correspond to subjects of either normal body weight, or obese, or suffering from lipodystrophic syndrome, whatever their type 2 diabetes status.

Methods: Blood IL-7 levels, other immune and/or pro-inflammatory cytokines, lymphocytes immuno-phenotype as well as metabolic parameters will be characterized. Fat mass will be assessed with non-invasive methods (DEXA and RMN). A plasma, serum and gene bank will be constituted. As well as an adipose tissue bank in patients who will have a surgery (especially plastic surgery in lipodystrophic patients), in order to cryo-preserve it and to define the inflammatory status of this tissue thanks to histological and molecular analysis.

Main judgment criteria: The main judgment criteria will be IL-7 blood levels in the different groups according to fat mass and metabolic parameters. The hypothesis is that in humans the quantitative and /or qualitative disturbances of adipose tissue are associated with an increase of IL-7 levels and the development of insulin-resistance.

Awaited results and possible implications: this study will allow to better delineate the immune and inflammatory component associated with alterations of fat mass distribution and glucose metabolism. Our approach combining clinical investigation and ex vivo and laboratory analysis is original and should allow to better understand the cellular mechanisms responsible for the inflammatory process originated in white adipose tissue and accompanying the disorders of this tissue- more especially lipodystrophic syndromes - opening new therapeutic perspectives in common human diseases (obesity, diabetes) on the one hand, and a rare disease (lipodystrophy) on the other hand.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* More than 18 years old
* with lipodystrophic syndrome (familial, partial, genetically determined), diabetics or not, obese or not
* Patients with lipodystrophy non related to a lamine A/C gene mutation, diabetics or not, obese or not
* Obese without diabetes (BMI> 30)
* Obese (BMI>30) and diabetes according to ADA criteria
* Normal weight patients (18< BMI< 25)
* Agreement for the establishment of a serum bank and a plasma bank

Exclusion Criteria:

* Unable to receive enlightened information
* Refusal to sign the consent
* Corticosteroids (including inhaled), other immunosuppressing treatments (systemic disease for example) or immunomodulators (eg interferon);
* Creatinin > 15 mg / L
* Sepsis
* Progressing cancers or autoimmune diseases;
* Treatment, disease or other condition that may affect the rate of IL-7 (as some contraceptives with estrogens)
* Bleeding disorders (due to disease or treatment)
* Active alcohol Intoxication
* Psychiatric pathology (after psychiatric consultation)
* Active infection including hepatitis C or HIV;
* Age under 18 years
* Participation in another study excluded the possibility of participating in another protocol
* BMI > 60
* Secondary diabetes
* No social security
* Pregnant or lactating women, patients under guardianship, persons deprived of liberty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with lipodystrophy : Endocrinology Departments of Lille , Amiens, Caen, Rouen and Reims University hospitals.
  Obese (diabetics and non diabetics) and normal weight patients : Endocrinology - Metabolism, Endocrine Surgery and Nutrition Departments, Lille University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2010-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measure of blood Interleukin 7 | 1 day

SECONDARY OUTCOMES:
measure of blood Interleukins 2 | 1 day
measure of blood interleukin 9 | 1 day
measure of blood Interleukin 15 | 1 day
measure of blood TNF | 1 day
measure of blood IL-1 | 1 day
measure of blood IL-6 | 1 day
measure of blood IL-8 | 1 day
measure of blood IL-10 | 1 day
measure of blood IL-18 | 1 day
measure of blood leptin | 1 day
measure of blood adiponectin | 1 day
Blood count of monocytes/macrophages | 1 day
Blood count of dendritic cells | 1 day
Count of blood lymphocytes T | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: marie christine VANTYGHEM, pHd, Principal Investigator — Lille University Hospital
Locations (5):
- France (5):
  - Amiens University Hospital, Amiens
  - Caen University Hospital, Caen
  - Lille University Hospital, Lille
  - Reims University Hospital, Reims
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemaitre M, Chevalier B, Jannin A, Le Mapihan K, Boury S, Lion G, Labalette M, Vantyghem MC. Metabolic and immunological phenotype of rare lipomatoses: Dercum's disease and Roch-Leri mesosomatic lipomatosis. Orphanet J Rare Dis. 2021 Jun 29;16(1):290. doi: 10.1186/s13023-021-01920-3. PMID 34187516